CLINICAL TRIAL: NCT06312488
Title: Point of Care Evaluation of Fibrinolysis in Sepsis
Acronym: POCEFIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Mauro Panigada, Principal Investigator, Policlinico Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4097
Record Dates: First submitted 2023-12-21; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Fibrinolytic Defect; Sepsis; Critical Illness
MeSH Terms: conditions — Fibrinolytic Defect; Sepsis; Critical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Septic patients (Other)
  Interventions: Diagnostic Test: Clot Pro
- Healthy volunteers (Other)
  Interventions: Diagnostic Test: Clot Pro

INTERVENTIONS:
Diagnostic Test: Clot Pro — This study enrolls patients admitted to the Adult ICU of Milan Policlinico Hospital with a diagnosis of sepsis or septic shock. A ClotPro® TPA test is performed at admission and on day 1, 2, 3, and 7. Specific markers of coagulation (PAI-1, Plasminogen, Protein C and S) and inflammation (Il-1beta, IL-6, IL-8, TNF-alpha, ADM) are tested at enrollment. Routine laboratory tests are performed daily. Hemorrhagic and thrombotic events are searched. The study ends at 28 days or upon ICU discharge.

SUMMARY:
Impaired fibrinolysis in septic patients is associated with worse outcome. The present study investigates fibrinolysis shutdown in septic patients, defined as prolonged ClotPro® TPA lysis time at 30 minutes. The TPA lysis time reference range is established in a cohort of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* sepsis or septic shock
* vasopressors required to maintain a MAP ≥ 65 mmHg despite adequate fluid resuscitation

Exclusion Criteria:

* coagulation disorders
* ECMO therapy
* use of oral anticoagulant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of impaired fibrinolysis | Lysis time at 30 minutes at enrollment and on day 1, 2, 3, and 7
  Lysis time at 30 minutes longer than 97.5th percentile of the calculated reference range of the ClotPro® TPA test

SECONDARY OUTCOMES:
Correlation between impaired fibrinolysis and changes in coagulation standard tests | Measures are performed at enrollment and on day 1, 2, 3, and 7
  Number of patients with impaired fibrinolysis who have other abnormalities in standard coagulation tests (increased PT and PTT, decreased platelet count, increased D-dimer and decreased fibrinogen)
Correlation between impaired fibrinolysis and inflammation markers | Measures are performed at enrollment and on day 1, 2, 3, and 7
  Number of patients with impaired fibrinolysis who have increased serum C-reactive protein and/or procalcitonin
Correlation between impaired fibrinolysis and multiorgan failure | Measures are performed at enrollment and on day 1, 2, 3, and 7
  Number of patients with impaired fibrinolysos who develop multiorgan failure, defined as SOFA score > 5
Correlation between impaired fibrinolysis and ICU lenght of stay | Through study completion, an average of 1 year
  Differential in number of days in ICU in patients with and without impaired fibrinolysis
Correlation between impaired fibrinolysis and ICU mortality | From date of enrollment until date of ICU discharge or date of death from any cause, whichever comes first, assessed up to 1 year
  Mortality rate in patients with and without impaired fibrinolysis

OTHER OUTCOMES:
Trend of fibrinolysis in the first ICU week with repeated ClotPro® tests | ClotPro® tests are performed at enrollment and on day 1, 2, 3, and 7
  Variation of TPA lysis time

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No